CLINICAL TRIAL: NCT04224077
Title: Optimisation of Diffusion Tensor Sequences (DTI) for Study of Lumbar Roots by Magnetic Resonance Imaging (MRI) : a Feasibility Study
Brief Title: Diffusion Tensor Sequences (DTI) for Study of Lumbar Roots by Magnetic Resonance Imaging (MRI)
Acronym: OPTI-DTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0060
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Radiculopathy Lumbar; MRI; Diffusion Tensor Imaging
Keywords: Radiculopathy Lumbar; MRI; Diffusion tensor imaging; Multiband technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Healthy volunteers
  Interventions: Diagnostic Test: Optimisation of DTI sequences

INTERVENTIONS:
Diagnostic Test: Optimisation of DTI sequences — Optimisation of DTI sequences in the study of lumbar roots by MRI

SUMMARY:
Diffusion tensor imaging (DTI) is a non-invasive MRI technique offering a functional approach that provides morphological information about the microstructures of the nerve roots. DTI is a widely used neuroimaging technique and is a current topic of research in the field of peripheral nerve imaging. The aim of this work is therefore to improve DTI sequences by specifically evaluating the contribution of the multiband technique in healthy volunteers.

DETAILED DESCRIPTION:
For every healthy volunteer will be acquired:

* a morphological sequence
* a reference diffusion tensor sequence covering three lumbar stages (reference DTI),
* a diffusion tensor sequence acquired in multiband technique, covering three lumbar stages (optimized DTI),
* a diffusion tensor sequence acquired in a multiband technique, covering a lumbar stage, of higher spatial resolution (centred DTI)

ELIGIBILITY:
Inclusion Criteria:

* Person without history of lumbar surgery
* Person who has previously consented

Exclusion Criteria:

* MRI contraindications (pace maker, cardiac defibrillator,...)
* Claustrophobia
* Pregnant woman
* Person without social security
* Person with a guardianship
* Person carrying metallic surgical material (spine, pelvis, abdomen)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Image quality measured as signal-to-noise ratio and contrast-to-noise ratio | Day 0
  Comparison of the image quality between DTI optimized and DTI of reference. The signal-to-noise ratio is a measure that compares the level of a desired signal to the level of background noise. Mathematically, the signal-to-noise ratio is the quotient of the (mean) signal intensity measured in a region of interest and the standard deviation of the signal intensity in a region outside the anatomy of the object being imaged.
  The contrast-to-noise ratio is a measure of image quality based on a contrast rather than the raw signal.

SECONDARY OUTCOMES:
Fraction of anisotropy and apparent diffusion coefficient | Day 0
  Comparison of fraction of anisotropy, and apparent diffusion coefficient between DTI optimized and DTI of reference.
  The measurement of fraction of anisotropy, and apparent diffusion coefficient provides robust values for quantifying the degree of microstructural abnormalities of nerves.
Concordance of observed agreement measured by Cohen's kappa coefficient | Day 0
  Evaluation of interobserver accordance for multiband acquisitions (optimized DTI)
Concordance of observed agreement measured by Intra-class correlation coefficient | Day 0
  Evaluation of interobserver accordance for multiband acquisitions (optimized DTI)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François BUDZIK, MD, Principal Investigator — GHICL
Locations (1):
- Lille Catholic Hospitals, Lomme, France

IPD SHARING:
Plan to Share IPD: No